CLINICAL TRIAL: NCT04534387
Title: Development and Assessment of a Spanish-Language Hearing Loss Toolkit for Self-Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21DC018655-01 (NIH); 1R21DC018655-01 (NIH)
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Self-Management; American Speech-Language-Hearing Association

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): This group will receive the Spanish-Language Hearing Loss Toolkit materials.
  Interventions: Other: Spanish-Language Hearing Loss Toolkit for Self-Management
- Active Control Group (Active Comparator): This group will receive standard of care Spanish language information from the American Speech-Language-Hearing Association (ASHA) Audiology Series
  Interventions: Other: American Speech-Language-Hearing Association (ASHA) Audiology Series Spanish Language Handouts

INTERVENTIONS:
Other: Spanish-Language Hearing Loss Toolkit for Self-Management — The materials include printed information and images designed to increase hearing loss knowledge and focus on self-management topics such as the fundamentals of the ear and hearing, communication strategies, speech understanding in noise, and hearing technology.
  Arms: Experimental Group
Other: American Speech-Language-Hearing Association (ASHA) Audiology Series Spanish Language Handouts — Standard of care patient education handouts developed by ASHA in the Spanish language.
  Arms: Active Control Group

SUMMARY:
The objective of this application is to develop and evaluate Spanish-language hearing education materials for adults. Our hypothesis is that participants will demonstrate better understanding of their hearing loss and associated difficulties, and will be better able to identify options for self-management following delivery of culturally and linguistically appropriate patient education materials.

DETAILED DESCRIPTION:
There are documented disparities in hearing healthcare use between Hispanic/Latino adults and non-Hispanic/Latino Whites, despite similar hearing loss prevalence rates. It has been suggested that a lack of culturally competent interventions contributes to poor healthcare delivery and outcomes for those with limited English proficiency. The objective of this application is to develop and evaluate Spanish-language hearing education materials for adults. Our hypothesis is that participants will demonstrate better understanding of their hearing loss and associated difficulties, and will be better able to identify options for self-management following delivery of culturally and linguistically appropriate patient education materials. The rationale for the proposed research is that findings will contribute to the development and testing of novel interventions aimed at increasing hearing healthcare access and utilization in vulnerable populations in a subsequent R01 application.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will include community-dwelling, Spanish-speaking (monolingual or bilingual) adults over age 50 who self-identify as Hispanic/Latino
2. Clinically-significant hearing loss defined as either greater than 25 decibels hearing leve (dB HL) thresholds at 2 or more frequencies from 250 - 8000 hertz (Hz) and/or significant self-reported hearing difficulties as defined by a score of greater than 8 on the Hearing Handicap Inventory - Screening measure for adults/elderly.

Exclusion Criteria:

* Individuals who are not fluent Spanish-speakers or who do not self-identify as Hispanic/Latino are not eligible to participate in this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Self-Efficacy for Hearing Loss Management (disease-specific primary outcome) | Assessed 4-6 weeks post baseline assessment
  Measured by the Partners in Health Scale-Audiology version. The original Partners in Health scale assesses management of chronic conditions and has been validated in several languages, including Spanish. Items are scored from 0-8 with higher scores indicating better self-management. The Partners in Health Scale-Audiology is an 11-item modified version of the original Partners in Health scale, and assesses the hearing loss-specific domains of actions, psychosocial behaviors, and knowledge.
Self-Efficacy for Chronic Health Condition Management (generic primary outcome) | Assessed 4-6 weeks post baseline assessment
  Measured by the Self-Efficacy to Mange Chronic Disease Scale-Spanish language version. The Self-Efficacy to Mange Chronic Disease Scale is a 4-item scale with high internal consistency (α=0.93) that measures changes in self-efficacy following participation in a disease self-management program. Items are scored from 1-10 with higher scores indicating better condition self-management.

SECONDARY OUTCOMES:
Hearing Loss Knowledge, Attitudes, and Behaviors | Assessed 4-6 weeks post baseline assessment
  Measured using the Hearing Beliefs Questionnaire. Assesses participants' knowledge, attitudes, and behaviors related to hearing loss at baseline and post-intervention. The Hearing Beliefs Questionnaire is a 26-item measure segmented into 6 domains: perceived susceptibility, perceived severity, perceived benefits, perceived barriers, perceived self-efficacy, and cues to action. Each domain includes between 3 and 8 visual analog scale items, with a range of adequate internal consistency of α=0.61-0.77. Possible score range for each item is 0 to 10, ranging from two endpoints of "highly agree" to "highly disagree" and "highly likely" to "highly unlikely". Item responses are averaged across domains as summary scores. As a Spanish-language version has not yet been validated, the Hearing Beliefs Questionnaire will be included as a secondary, exploratory outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Arnold, Au.D., Ph.D., Principal Investigator — University of South Florida; Victoria Sanchez, Au.D., Ph.D., Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available upon the close of the study (March 30, 2023) and will remain available for 1 year post study-closure (March 30, 2024).
Access Criteria: Individuals requesting access must meet qualifications for Institution and Investigator detailed in the National Institute on Deafness and Other Communication Disorders (NIDCD) Funding Opportunity Announcement Number described in PAR-18-487.

DOCUMENTS (1):
  • Informed Consent Form (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT04534387/ICF_000.pdf